CLINICAL TRIAL: NCT06497699
Title: A Real-world Study to Evaluate the Efficacy and Safety of 9% Dexamethasone Intraocular Injection for the Treatment of Inflammation Associated With Cataract Surgery
Brief Title: A Real-world Study of DEXYCU in the Treatment of Inflammation After Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ocumension Therapeutics (Shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Ocumension Therapeutics (Suzhou) Co., Ltd (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OT-502-002
Record Dates: First submitted 2024-06-20; First posted 2024-07-12 (Actual); Results first posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Inflammation; Cataract
Keywords: Cataract Surgery; Postoperative Inflammation
MeSH Terms: conditions — Inflammation; Cataract | interventions — Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: Study group:Dexycu interventional group
  External control group;without intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study Group (Experimental): Single injection of DEXYCU in the treatment eye after cataract surgery.
  Interventions: Drug: Dexycu
- Control Group (No Intervention): The clinical routine treatment after cataract surgery was adopted without intervention

INTERVENTIONS:
Drug: Dexycu — single injection,5ul solution,concentration: 103.4 μg/μl, equivalent to 517μg dexamethasone
  Arms: Study Group

SUMMARY:
This is a prospective, real-world study aimed to evaluate the efficacy and safety of Dexycu in treating postoperative inflammation of cataracts.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of Dexycu in treating postoperative inflammation of cataracts in real-world clinical settings, medical history and follow-up data from 113 subjects of Dexycu group and 150 subjects of external control group will be prospectively collected in Hainan, China. Additionally, questionnaires will be collected from surgeons on 30 cases to evaluate the difficulty, duration and safety of the Dexycu injector.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to understand and sign the informed consent form and be able to follow the study procedures.
* Male or female subjects over 40 years of age who are scheduled to undergo cataract phacoemulsification surgery combined with intraocular lens implantation.

Exclusion Criteria:

* Known hypersensitivity to dexamethasone or any component of the Dexycu.
* History of intraocular inflammation of any cause in either eye, presence of corneal abnormalities or malnutrition.
* Have high intraocular pressure, with an IOP(intraocular pressure) of > 21 mmHg in the test eye at screening, regardless of whether receiving anti-glaucoma monotherapy therapy.
* Posterior capsule rupture or lens dislocation, anterior vitreal membrane rupture, vitreous prolapse and intraoperative floppy iris syndrome during cataract surgery.
* Other conditions that the investigator considers inappropriate to participate the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2023-07-08 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhixun Li, Study Director — Ocumension Therapeutics (Shanghai) Co., Ltd
Locations (2):
- China (2):
  - Hainan Traditional Chinese Medicine Hospital, Haikou, Hainan
  - Boao Super Hospital, Bo'ao

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 113 recruited to the study group treat with DEXYCU postsurgerically. 150 recruited to control group which observation study was conducted.
Units Other Than Participants: Eye
Period: Overall Study
Arm/Group | Control Group | Study Group
Started | 150; 150 Eye | 113; 113 Eye
Completed | 143; 143 Eye | 110; 110 Eye
Not Completed | 7; 7 Eye | 3; 3 Eye

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Study Group | Total
Number analyzed (Participants) | 150 | 113 | 263
Age, Customized [Count of Participants; unit: Participants]
  < = 60 years | 15 | 17 | 32
  > 60 years | 135 | 96 | 231
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 55 | 139
  Male | 66 | 58 | 124
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 150 | 113 | 263
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 149 | 113 | 262

OUTCOME MEASURES:

1. Primary Outcome: Anterior Chamber Cell Clearing Rate
Description: The primary outcome is to compare the ratio of subjects with anterior chamber cell grade 0 at day 8 after cataract surgery of both Dexycu group and external control group.
  The slit lamp examination for anterior chamber cells (ACC) is a recognized way to measure inflammation in the anterior chamber. During the slit lamp examination, the number of anterior chamber cells are quantified and graded: grade 0 (absent, 0 cells), grade 1 (1 to 5 cells), grade 2 (6 to 15 cells), grade 3 (16 to 30+ cells), or grade 4 (hypopyon). Anterior chamber cell clearing occurs when all the ACC are absent (grade 0).
Time Frame: DAY 8
Population: 1 control group participant loss to follow up before reaching DAY 8.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 149 | 113
Participants | 119 | 95

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 90 days
Arm/Group | Control Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/150 | 1/113
Serious Adverse Events (participants affected / at risk) | 5/150 | 1/113
Other Adverse Events (participants affected / at risk) | 14/150 | 15/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=150) | Study Group (N=113)
Endophthalmitis (Eye disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Macular Oedema (Eye disorders) | 4 (4) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=150) | Study Group (N=113)
Corneal endothelial cell loss (Eye disorders) | 14 (14) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT06497699/Prot_SAP_000.pdf